CLINICAL TRIAL: NCT02151149
Title: Safety and Efficacy of Nab-paclitaxel (Abraxane) in Combination With Carboplatin as First Line Treatment in Elderly Subjects With Advance Non-Small Cell Lung Cancer (NSCLC): A Phase IV, Randomized, Open-Label, Multicenter Study (Abound.70+)
Brief Title: Safety and Efficacy Study of Abraxane in Combination With Carboplatin to Treat Advanced NSCL Cancer in the Elderly
Acronym: ABOUND 70+
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABI-007-NSCL-005
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Results first posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-08

CONDITIONS: Non-Small Cell Lung Cancer; Carcinoma; Squamous Cell Carcinoma; Adenocarcinoma; Carcinoma, Large Cell; Lung Neoplasm
Keywords: NSCLC advanced non-small cell lung cancer squamous adenocarcinoma large cell carcinoma lung cancer elderly first line treatment abraxane carbo nab-paclitaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma; Carcinoma, Squamous Cell; Adenocarcinoma; Carcinoma, Large Cell; Lung Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: nab-Paclitaxel and Carboplatin (Every 21 days) (Other): nab-Paclitaxel 100 mg/m2 intravenous (IV) infusion over 30 minutes on Days 1, 8, and 15 and Carboplatin AUC = 6 mg*min/mL IV following nab-paclitaxel infusion on Day 1 of every 21-day treatment cycle
  Interventions: Drug: nab-paclitaxel; Drug: Carboplatin
- Arm B: nab-Paclitaxel and Carboplatin (Every 28 days) (Other): nab-Paclitaxel 100 mg/m2 IV infusion over 30 minutes on Days 1, 8, and 15 of each 21-day treatment followed by one-week break and Carboplatin AUC = 6 mg*min/mL IV following nab-paclitaxel infusion on Day 1 of each 21-day treatment followed by one-week break
  Interventions: Drug: nab-paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: nab-paclitaxel
  Other Names: Abraxane
Drug: Carboplatin

SUMMARY:
Study comparing two regimens of nab-paclitaxel and carboplatin combination in elderly subjects (≥ 70 years old) with advanced NSCLC

DETAILED DESCRIPTION:
This is a Phase IV, randomized, open-label, multicenter study of continuous weekly versus weekly times three with one-week break nab-paclitaxel in combination with carboplatin as first-line treatment in elderly subjects (≥ 70 years old) with advanced non small cell lung cancer who have not received prior chemotherapy for their advanced disease and are not candidates for curative surgery or radiation therapy. The primary study endpoint is the percentage of subjects with either peripheral neuropathy or myelosuppression adverse events. Patients will continue treatment until they develop progressive disease, unacceptable side-effects or wish to withdraw from the study, according to local standard of care. Patients will have radiographic evaluations every 6 weeks while on treatment.

ELIGIBILITY:
Inclusion Criteria: -

* Inclusion Criteria: -

  1. Age ≥ 70 years at the time of signing the Informed Consent Form.
  2. Understand and voluntarily provide written informed consent prior to the conduct of any study related assessments/procedures.
  3. Able to adhere to the study visit schedule and other protocol requirements.
  4. Histologically or cytologically confirmed locally advanced or metastatic non small cell lung cancer who are not candidates for curative surgery or radiation therapy.
  5. No other current active malignancy requiring anticancer therapy.
  6. Radiographically documented measurable disease per RECIST v 1.1
  7. No prior chemotherapy for the treatment of metastatic disease. Adjuvant chemotherapy is permitted providing that cytotoxic chemotherapy was completed 12 months prior to signing the informed consent form (ICF) and without disease recurrence. Participans with previously known epidermal growth factor receptor mutation or anaplastic lymphoma kinase gene translocation must have failed or had intolerance to one treatment with epidermal growth factor receptor tyrosine kinase inhibitor or anaplastic lymphoma kinase inhibitor therapy, respectively.
  8. Absolute neutrophil count ≥ 1500 cells/cubic millimetre.
  9. Platelets ≥ 100,000 cells/cubic millimetre.
  10. Hemoglobin ≥ 9 grams/decilitre.
  11. Aspartate transaminase/serum glutamic oxaloacetic transaminase/ alanine transaminase/serum glutamic pyruvic transaminase ≤ 2.5 × upper limit of normal range or ≤ 5.0 × upper limit of normal range if liver metastases.
  12. Total bilirubin ≤ 1.5 millilitre/decilitre (unless there is a known history of Gilberts Syndrome).
  13. Creatinine clearance > 40 millilitre/minute calculated using Cockcroft-Gault equation (if renal impairment is suspected 24 hour urine collection for measurement is required).
  14. Eastern Cooperative Oncology Group performance status 0 or 1.
  15. Females who (1) have undergone hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or (2) have been naturally postmenopausal for at least 24 consecutive months (ie, has not had menses at any time during the preceding 24 consecutive months).
  16. Male subjects must: Practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for 6 months following study drug discontinuation, even if he has undergone a successful vasectomy.

      Exclusion Criteria:
* 1. Evidence of active brain metastases, including leptomeningeal involvement (prior evidence of brain metastasis are permitted only if treated and stable and off therapy for ≥ 4 weeks prior to signing Informed consent form. Magnetic Resonance Imaging of the brain (or Computed Tomography scan w/contrast) is preferred for diagnosis.

  2. History of leptomeningeal disease. 3. Only evidence of disease is non measurable. 4. Preexisting peripheral neuropathy of Grade 2, 3, or 4 (per Common Terminology Criteria for Adverse Events v4.0).

  5. Participant has received radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting investigational product, and/or from whom ≥ 30% of the bone marrow was irradiated. Prior radiation therapy to a target lesion is permitted only if there has been clear progression of the lesion since radiation was completed.

  6. Venous thromboembolism within 1 month prior to signing informed consent form.

  7. Current congestive heart failure (New York Heart Association Class II-IV). 8. History of the following within 6 months prior to first administration of a study drug: a myocardial infarction, severe/unstable angina pectoris,coronary/peripheral artery bypass graft, New York Heart Association Class III-IV heart failure, uncontrolled hypertension, clinically significant cardiac dysrhythmia or clinically significant Electrocardiogram abnormality, cerebrovascular accident, transient ischemic attack, or seizure disorder.

  9. Participant has a known infection with hepatitis B or C, or history of human immunodeficiency virus infection, or participant is receiving immunosuppressive or myelosuppressive medications that would in the opinion of the investigator, increase the risk of serious neutropenic complications.

  10. Participant has an active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy, defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment.

  11.History of interstitial lung disease, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, or pulmonary hypersensitivity pneumonitis.

  12. Treatment with any investigational product within 28 days prior to signing the informed consent form.

  13. History of allergy or hypersensitivity to nab-paclitaxel or carboplatin. 14. Currently enrolled in any other clinical protocol or investigational trial that involves administration of experimental therapy and/or therapeutic devices. 15. Any other clinically significant medical condition, psychiatric illness, and/or organ dysfunction that will interfere with the administration of the therapy according to this protocol or which, in the views of investigator, preclude combination chemotherapy.

  16. Participant has any other malignancy within 5 years prior to randomization. Exceptions include the following: squamous cell carcinoma of the skin, in-situ carcinoma of the cervix, uteri, non-melanomatous skin cancer, carcinoma in situ of the breast, or incidental histological finding of prostate cancer Tumor, Lymph Node, Metastatic (TNM stage of T1a or T1b). All treatment of which should have been completed 6 months prior to signing Informed consent form.

  17. Any condition including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study.

  18. Any medical condition that confounds the ability to interpret data from the study.

  19. Females who (1) have not undergone hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or (2) have not been naturally postmenopausal for at least 24 consecutive months (ie, has had menses at any time during the preceding 24 consecutive months).

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 143 (Actual)
Dates: Start 2014-06-09 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teng Jin Ong, Study Director — Celgene
Locations (55):
- United States (55):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Saint Jude Heritage Medical Center, Fullerton, California
  - Global Cancer Research Institute (GCRI), Inc., Gilroy, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - University of California Los Angeles, Santa Monica, California
  - Rocky Mountain Cancer Centers, LLP, Denver, Colorado
  - St Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Lynn Cancer Institute, Boca Raton, Florida
  - Baptist Cancer Inst, Jacksonville, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Northshore University Healthsystem Research Institute, Evanston, Illinois
  - Oncology Specialists, S.C., Niles, Illinois
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Western Kentucky Hematology and Oncology Group, Paducah, Kentucky
  - West Jeffersion Medical Center, Marrero, Louisiana
  - Ochsner Medical Institutions, New Orleans, Louisiana
  - Medstar Health Research Institute, Baltimore, Maryland
  - Reliant Medical Group, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - Regional Cancer Care Associates LLC, East Brunswick, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Carol G Simon Cancer Center, Morristown, New Jersey
  - Somerset Hematology-Oncology Associates, Somerville, New Jersey
  - Regional Cancer Care Associates LLC- Sparta division, Sparta, New Jersey
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Broome Oncology, LLC, Johnson City, New York
  - Clinical Research Alliance, Lake Success, New York
  - SUNY Upstate Medical University Medicine Oncology, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Lineberger Cancer Center, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Forsyth Memorial Hospital, Inc., Winston-Salem, North Carolina
  - St Elizabeth Hospital, Youngstown, Ohio
  - Cancer Centres of Southwest Okahoma Research, Lawton, Oklahoma
  - Good Samaritan Hospital Corvalis, Corvallis, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University Medical College, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Texas Oncology, P.A.-Amarillo, Amarillo, Texas
  - Baylor University Medical Center at Dallas, Dallas, Texas
  - UTMB Galveston, Galveston, Texas
  - Texas Oncology, PA - Longview, Longview, Texas
  - Virginia Mason Cancer Center, Seattle, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in the United States and enrolled participants at a total of 41 sites.
Pre-assignment Details: Participants ≥ 70 years old were randomized 1:1 to nab-paclitaxel and carboplatin on a 21-day treatment regimen or nab-paclitaxel and carboplatin on a 28-day treatment regimen; participants were stratified by Eastern Cooperative Oncology Group performance status (0 versus 1) and histology (squamous cell carcinoma versus non-squamous cell carcinoma)
Groups:
- Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce): Participants ≥ 70 years old received nab-paclitaxel 100 mg/m^2 by intravenous (IV) infusion over 30 minutes on Days 1, 8, and 15 of each 21-day treatment cycle and carboplatin area under the curve (AUC) at 6 mg*min/mL IV on Day 1 of each 21-day cycle after completion of nab-paclitaxel infusion until disease progression, development of an unacceptable toxicity, death, lost to follow-up, or withdrawal of consent, in accordance with local standard of care.
- Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle): Participants ≥ 70 years old received nab-paclitaxel 100 mg/m^2 by intravenous infusion over 30 minutes on Days 1, 8, and 15 followed by a one-week break in each 28-day treatment cycle and carboplatin area under the curve of 6 mg*min/mL IV on Day 1 after completion of nab-paclitaxel infusion of each treatment cycle until disease progression, development of an unacceptable toxicity, death, lost to follow-up, or withdrawal of consent, in accordance with local standard of care.
Period: Treatment Period
Arm/Group | Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) | Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle)
Started | 71 (3 participants did not receive treatment) | 72 (2 participants did not receive treatment)
Treated Population | 68 | 70
Completed (Completed indicates participants with missing disposition data.) | 1 | 1
Not Completed | 70 | 71
Not completed — Death | 2 | 3
Not completed — Adverse Event | 17 | 14
Not completed — Progressive Disease | 25 | 24
Not completed — Symptomatic Deterioration | 2 | 10
Not completed — Withdrawal by Subject | 13 | 11
Not completed — Miscellaneous | 8 | 7
Not completed — Participants randomized but not treated | 3 | 2
Period: Follow-Up Period
Arm/Group | Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) | Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle)
Started | 58 | 55
Completed | 19 (Completed = participants alive at final data cut-off date) | 18 (Completed = participants alive at final data cut-off date)
Not Completed | 39 | 37
Not completed — Lost to Follow-up | 2 | 3
Not completed — Death | 37 | 34

BASELINE CHARACTERISTICS:
Population: Intent to Treat Population included all randomized participants regardless of whether the participant received any study drug or had any efficacy assessments performed.
Groups:
- Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle): Participant ≥ 70 years old received nab-paclitaxel 100 mg/m^2 by intravenous infusion over 30 minutes on Days 1, 8 and 15 followed by a one week break in each 28-day treatment cycle and carboplatin area under the curve (AUC) = 6 mg*min/mL IV on Day 1 of each treatment cycle after completion of nab-paclitaxel infusion until disease progression, development of an unacceptable toxicity, death, lost to follow-up, or withdrawal of consent, in accordance with local standard of care.
- Total: Total of all reporting groups
Arm/Group | Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) | Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle) | Total
Number analyzed (Participants) | 71 | 72 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.7 (4.13) | 76.4 (5.18) | 76.6 (4.67)
Age, Customized [Count of Participants; unit: Participants]
  70-74 years | 20 | 33 | 53
  75-79 years | 30 | 18 | 48
  80-84 years | 19 | 17 | 36
  85-89 years | 2 | 2 | 4
  ≥ 90 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 62
  Male | 41 | 40 | 81
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 3 | 3
  Black or African American | 3 | 7 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 64 | 57 | 121
  Other | 1 | 1 | 2
  Data Missing | 3 | 2 | 5
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Number; unit: Participants] — ECOG performance status is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity)
  Participants
    0 = Fully Active | 21 | 20 | 41
    1 = Restricted in Physical Activity; Ambulatory | 50 | 52 | 102
    2 = Ambulatory and Capable of All Self-care | 0 | 0 | 0
    3 = Capable of Only Limited Self-care | 0 | 0 | 0
    4 = Completely Disabled. | 0 | 0 | 0
Confirmed Histology [Count of Participants; unit: Participants]
  Squamous Cell Carcinoma | 27 | 28 | 55
  Non-Squamous Cell Carcinoma | 44 | 44 | 88
Stage of Disease at Enrollment [Count of Participants; unit: Participants] — Disease stage means how big the tumor is and how far it has spread. Disease stages range from 0 (not spread) to IV (spread throughout the body). Stage III - the cancer has spread to nearby tissue or spread to far away lymph nodes; if the tumor has spread only to the lymph nodes on the same side of the chest where the cancer started, it is Stage IIIA; if the tumor has spread to the lymph nodes on the opposite side or above the collar bone, it is Stage IIIb. Stage IV - the cancer has spread to other organs of the body such as the other lung, brain, or liver.
  Participants
    IIIa | 4 | 5 | 9
    IIIb | 6 | 8 | 14
    IV | 60 | 59 | 119
    Data Missing | 1 | 0 | 1
Number of Prior Systemic Anticancer Therapies for Non-Small Cell Lung Cancer (NSCLC) [Median (Full Range); unit: Therapies] | 2.0 [1.0 to 2.0] | 2.0 [2.0 to 4.0] | 2.0 [1.0 to 4.0]
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] — Body Mass Index = (Weight in kg) / (Height in m)^2. Population: 1 participant's disposition is missing
  Kg/m^2
    number analyzed (Participants) | 70 | 72 | 142
    (all) | 26.357 (4.6805) | 26.033 (4.7562) | 26.193 (4.7051)
Number of Participants with Peripheral Neuropathy at Baseline [Count of Participants; unit: Participants] — Physician assessment for grading of peripheral neuropathy in participants receiving chemotherapy according to National Cancer Institute Common Toxicity Criteria (NCICTC):
  Grade 1 = Asymptomatic: loss of deep tendon reflexes or paresthesia; Grade 2 = Moderate symptoms: limiting instrumental Activities of Daily Living (ADLs); Grade 3 = Severe symptoms: limiting self-care ADL; assistance device indicated; Grade 4 = Life-threatening consequences: urgent intervention indicated.
  Participants
    No Peripheral Neuropathy | 54 | 57 | 111
    Grade 1 | 14 | 13 | 27
    Grade 2 | 1 | 0 | 1
    Data Missing | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Either Peripheral Neuropathy ≥ Grade 2 or Myelosuppression Adverse Events (AEs) ≥ Grade 3 Based on Local Laboratory Values
Description: Peripheral neuropathy (sensory or motor) assessment was done at screening, on Days 1, 8, 15 of every treatment cycle, at the End-of-Treatment visit and at the 28-day Follow-up Visit. Changes in neuropathy grade from baseline was reported as an AE as assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0. Myelosuppression in participants receiving chemotherapy may have manifested as neutropenia, thrombocytopenia, or anemia. Grade 3 neutropenia including an absolute neutropenia count (ANC) of 500 to 1,000 cells/mm^3; anemia hemoglobain levels (Hgb) <8.0 - 6.5 g/dL; <4.9 - 4.0 mmol/L; <80 - 65 g/L; transfusion indicated; and thrombocytopenia with platelet levels <100,000 cells/mm^3.
Time Frame: From the date of the first dose of investigational product (IP) until 28 days after the last dose of IP; up to data cut-off date of 20 November 2016; The median treatment duration for Arms A and B were 3.04 months and 5.17 months respectively.
Population: Treated Population included all participants who were randomized and received at least 1 dose of the study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) | Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle)
Number analyzed (Participants) | 68 | 70
Percentage of Participants | 76.5 [64.6 to 85.9] | 77.1 [65.6 to 86.3]
Statistical Analysis 1: Comparison: Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) vs Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle); Test type: Superiority; p = 0.9258, Cochran-Mantel-Haenszel; Based on stratification factors of ECOG PS at screening (0 vs. 1) and histology (squamous cell carcinoma vs. non-squamous cell carcinoma); Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.84 to 1.21]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events During the Treatment Period
Description: Treatment-emergent adverse events (TEAEs) were defined as any AE or serious adverse event (SAE) that occurred or worsened on or after the day of the first dose of the IP through 28 days after the last dose of IP. Any SAE with an onset date more than 28 day after the last dose of IP that was assessed by the investigator as related to IP was considered a TEAE. The severity of AEs was graded based on National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0 and based on the scale:
  Grade 1 = Mild - transient or mild discomfort; Grade 2 = Moderate - mild to moderate limitation in activity, assistance may be needed; minimal medical intervention required; Grade 3 = Severe - marked limitation in activity, assistance usually required; medical intervention required, hospitalization is possible; Grade 4 = Life threatening - extreme limitation in activity, assistance required; medical intervention, hospitalization or hospice care probable; Grade 5 = death.
Time Frame: From the date of the first dose of IP until 28 days after the last dose of IP; up to a later data cut-off date of 14 July 2017; maximum treatment duration for Arms A and B was 16.6 months and 20.1 months respectively.
Population: Safety population included all participants who were randomized and received at least 1 dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) | Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle)
Number analyzed (Participants) | 68 | 70
Participants
  Treatment Emergent Adverse Event | 68 | 69
  Serious Treatment Emergent Adverse Event | 23 | 32
  Grade 3 or 4 Treatment Emergent Adverse Event | 60 | 59
  Grade 3 or Higher Treatment Emergent Adverse Event | 60 | 61
  Treatment Related TEAE | 65 | 66
  Treatment-Related Serious TEAE | 12 | 12
  TEAE with Action to Reduce or Interrupt IP Dose | 60 | 54
  Treatment-Related Action to Reduce/Interrupt IP | 56 | 51
  TEAE with Action Taken as Study Drug Withdrawn | 17 | 14
  Treatment-related TEAE with Action to Halt IP | 13 | 13
  TEAE with Fatal Outcome | 1 | 3
  Treatment-related TEAE with Fatal Outcome | 0 | 0

3. Secondary Outcome: Percentage of Participants With at Least 1 Treatment Emergent Adverse Event With Action Taken as Study Drug Withdrawn
Description: The percentage of participants with at least 1 TEAE with action taken as studydrug withdrawn during the treatment period of the trial was assessed throughout the conduct of the study. Study drug withdrawn (treatment permanently discontinued) was attributed to the part in which the onset of the adverse event took place.
Time Frame: From the date of the first dose of IP until 28 days after the last dose of IP; up to a later data cut-off date of 14 July 2017 the maximum treatment duration for Arms A and B was 16.6 months and 20.1 months respectively
Population: Safety Population included all participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) | Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle)
Number analyzed (Participants) | 68 | 70
Percentage of Participants | 25.0 | 20.0

4. Secondary Outcome: Dose Intensity Per Week of Nab-Paclitaxel During the Entire Study
Description: Dose intensity was the cumulative dose divided by the dosing period in weeks.
Time Frame: From day 1 of study treatment to the end date of study treatment; up to data cut off date of 20 November 2016; the maximum treatment duration for Arms A and B was 16.6 months and 20.1 months respectively
Population: Treated Population included all randomized participants who received any study drug.
Measure: Mean (Standard Deviation); unit: mg/m^2/week
Arm/Group | Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) | Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle)
Number analyzed (Participants) | 68 | 70
mg/m^2/week | 64.07 (17.374) | 56.57 (16.645)

5. Secondary Outcome: Dose Intensity Per Week of Carboplatin During the Entire Study
Description: Dose intensity for carboplatin was the cumulative dose divided by the dosing period in weeks."
Time Frame: as for outcome 4
Population: Treated Population included all randomized participants who received any study drug.
Measure: Mean (Standard Deviation); unit: mg*min/mL/week
Arm/Group | Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) | Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle)
Number analyzed (Participants) | 68 | 70
mg*min/mL/week | 1.51 (0.384) | 1.33 (0.671)

6. Secondary Outcome: Percentage of Participants With Dose Reductions During the Entire Study
Description: A dose reduction occurred when the dose assigned at a visit was lower than the dose assigned at the previous visit. Dose reductions were typically caused by clinically significant laboratory abnormalities and/or TEAEs or toxicities.
Time Frame: From the first dose of study treatment to discontinuation date of study treatment; up to date cut off date of 20 November 2016; the maximum treatment duration for Arms A and B was 16.6 months and 20.1 months respectively
Population: The treated population consisted of all participants who received at least 1 dose of investigational product.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) | Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle)
Number analyzed (Participants) | 68 | 70
Percentage of Participants
  nab-Paclitaxel | 64.7 | 58.6
  Carboplatin | 57.4 | 58.6

7. Secondary Outcome: Percentage of Participants With a Dose Delay During the Entire Study
Description: A dose delay occurred when the dose assigned at a visit was held compared to the previous visit. Dose delays were typically caused by clinically significant laboratory abnormalities and/or TEAEs or toxicities.
Time Frame: From the first dose of study treatment to discontinuation date of study treatment; up to date cut off date of 16 November 2016; the maximum treatment duration for Arms A and B was 16.6 months and 20.1 months respectively
Population: The safety population consisted of all participants who received at least 1 dose of investigational product.
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) | Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle)
Number analyzed (Participants) | 68 | 70
Percentage of Participants
  nab-Paclitaxel | 58.8 | 48.6
  Carboplatin | 52.9 | 44.3

8. Secondary Outcome: Kaplan Meier Estimate of Progression-Free Survival (PFS)
Description: Progression-free survival was defined as the time in months from day 1 of treatment to the date of disease progression based on the investigator's assessment according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 criteria (documented by radiological assessment) or death (any cause) on or prior to the clinical cut-off date, which ever occurred earlier. RECIST V1.1 criteria includes: - Complete Response (CR) is the disappearance of all target lesions; - Partial Response (PR) is at least a 30% decrease in the sum of diameters of target lesions from baseline; - Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase of lesions to qualify for progressive disease (PD); - Progressive Disease is at least a 20% increase in the sum of diameters of target lesions from nadir
Time Frame: From first dose of IP to the date of disease progression; up to a later clinical cut-off date of 14 July 2017; for Arms A and B participants were followed for PFS for 31 months and 20 months respectively
Population: Intent to Treat Population all randomized participants regardless of whether the participant received any study drug or had any efficacy assessments performed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) | Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle)
Number analyzed (Participants) | 71 | 72
months | 3.88 [3.02 to 6.24] | 7.20 [5.85 to 11.53]
Statistical Analysis 1: Comparison: Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) vs Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle); Test type: Superiority; p = 0.0036, Stratified Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.33 to 0.81]

9. Secondary Outcome: Kaplan Meier Estimate of Overall Survival (OS)
Description: Overall survival was defined as the time in months between day 1 of treatment and death from any cause). Participants who were still alive as of the clinical cut-off date had their OS censored at the date of last contact or clinical cut-off, whichever was earlier. Participants who were lost to follow-up prior to the end of the study or who were withdrawn from the study were censored at the time of last contact.
Time Frame: From first dose of IP to the date of death due to any cause; up to a later clinical cut-off date of 14 July 2017; for Arms A and B participants were followed for OS for 31 months and 33 months respectively
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) | Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle)
Number analyzed (Participants) | 71 | 72
months | 14.52 [9.46 to 17.28] | 14.98 [12.09 to 18.73]
Statistical Analysis 1: Comparison: Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) vs Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle); Test type: Superiority; p = 0.3537, Stratified log-rank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.54 to 1.25]

10. Secondary Outcome: Percentage of Participants Who Achieved a Best Overall Response of Complete Response (CR) or Partial Response (PR) According to RECIST 1.1 Criteria
Description: Overall response rate (ORR) was defined as the percentage of participants who had radiologic CR or PR compared to baseline (radiographic evaluation on the day of or within 28 days prior to randomization) according to RECIST Version 1.1 criteria as determined by the investigator, which was confirmed by repeated radiologic assessment performed no less than 28 days after the criteria for response were first met and occurred between Day 1 of treatment and the start of subsequent anticancer therapy, death or study discontinuation. A complete response and partial response per RECIST V 1.0 criteria was defined as the disappearance of all target lesions; a partial response was defined as at least a 30% decrease in the sum of diameters of target lesions from baseline.
Time Frame: From the first dose of IP to the date of documented first response; up to the data cut-off date of 14 July 2017; maximum treatment duration for Arms A and B was 16.6 months and 20.1 months respectively.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) | Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle)
Number analyzed (Participants) | 71 | 72
Percentage of participants | 26.8 [16.9 to 38.6] | 41.7 [30.2 to 53.9]
Statistical Analysis 1: Comparison: Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) vs Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle); Test type: Superiority; p = 0.0597, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.56, 95% CI 2-sided [0.971 to 2.511]

ADVERSE EVENTS:
Time Frame: TEAEs are reported up to 37 months; from Day 1 of IP until 28 days after the last dose of IP and those SAEs made known to the Investigator at any time thereafter being suspected of being related to IP; up data cut-off date of 14 July 2017.
Arm/Group | Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) | Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle)
All-Cause Mortality (participants affected / at risk) | 45/71 | 46/72
Serious Adverse Events (participants affected / at risk) | 23/68 | 32/70
Other Adverse Events (participants affected / at risk) | 68/68 | 69/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) (N=68) | Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle) (N=70)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 3
Atrial flutter (Cardiac disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Gallbladder obstruction (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 5
Sepsis (Infections and infestations) | 1 | 0
Serratia infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 2
Delirium (Psychiatric disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nab-Paclitaxel and Carboplatin (21-day Treatment Cylce) (N=68) | Arm B: Nab-Paclitaxel and Carboplatin (28-day Treatment Cycle) (N=70)
Anaemia (Blood and lymphatic system disorders) | 45 | 39
Leukopenia (Blood and lymphatic system disorders) | 14 | 11
Neutropenia (Blood and lymphatic system disorders) | 35 | 32
Thrombocytopenia (Blood and lymphatic system disorders) | 30 | 19
Vision blurred (Eye disorders) | 3 | 4
Abdominal pain (Gastrointestinal disorders) | 9 | 9
Constipation (Gastrointestinal disorders) | 25 | 20
Diarrhoea (Gastrointestinal disorders) | 29 | 26
Dysphagia (Gastrointestinal disorders) | 4 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 6
Nausea (Gastrointestinal disorders) | 32 | 37
Stomatitis (Gastrointestinal disorders) | 14 | 8
Vomiting (Gastrointestinal disorders) | 13 | 20
Asthenia (General disorders) | 7 | 3
Chills (General disorders) | 1 | 6
Fatigue (General disorders) | 46 | 37
Non-cardiac chest pain (General disorders) | 3 | 5
Oedema peripheral (General disorders) | 12 | 13
Pain (General disorders) | 6 | 1
Pyrexia (General disorders) | 5 | 7
Oral candidiasis (Infections and infestations) | 4 | 0
Pneumonia (Infections and infestations) | 4 | 5
Upper respiratory tract infection (Infections and infestations) | 6 | 3
Urinary tract infection (Infections and infestations) | 7 | 6
Contusion (Injury, poisoning and procedural complications) | 4 | 1
Fall (Injury, poisoning and procedural complications) | 5 | 7
Overdose (Injury, poisoning and procedural complications) | 6 | 1
Blood creatinine increased (Investigations) | 1 | 4
Neutrophil count decreased (Investigations) | 14 | 13
Platelet count decreased (Investigations) | 9 | 6
Weight decreased (Investigations) | 9 | 13
White blood cell count decreased (Investigations) | 5 | 7
Decreased appetite (Metabolism and nutrition disorders) | 22 | 26
Dehydration (Metabolism and nutrition disorders) | 16 | 17
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 17
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 14
Hyponatraemia (Metabolism and nutrition disorders) | 11 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 7
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 13
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 8
Dizziness (Nervous system disorders) | 14 | 14
Dysgeusia (Nervous system disorders) | 7 | 10
Headache (Nervous system disorders) | 7 | 7
Peripheral motor neuropathy (Nervous system disorders) | 7 | 11
Peripheral sensory neuropathy (Nervous system disorders) | 40 | 30
Anxiety (Psychiatric disorders) | 2 | 10
Insomnia (Psychiatric disorders) | 8 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 | 10
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 27 | 29
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 | 8
Hypertension (Vascular disorders) | 1 | 4
Hypotension (Vascular disorders) | 4 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than one year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to ninety days. Investigator must delete confidential information before submission or defer publication to permit patent applications

DOCUMENTS (6):
  • Statistical Analysis Plan: ABI-007-NSCL-005_SAP_AM!_Redacted.17March 2016 (2016-03-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT02151149/SAP_000.pdf
  • Study Protocol: ABI-007-NSCL-005_PA1_Redacted.09April2014 (2014-04-09): https://cdn.clinicaltrials.gov/large-docs/49/NCT02151149/Prot_001.pdf
  • Statistical Analysis Plan: ABI-007-NSCL-005.OriginalSAP.Redacted24 June2016 (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/49/NCT02151149/SAP_002.pdf
  • Study Protocol: ABI-007-NSCL-005_PA2_Redacted.05 December 2014 (2014-12-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT02151149/Prot_003.pdf
  • Study Protocol: ABI-007-NSCL-005_PA3_Redacted.17 March 2016 (2016-03-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT02151149/Prot_004.pdf
  • Study Protocol: ABI-007-NSCL-005_Original_Redacted.06 March2014 (2014-03-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT02151149/Prot_005.pdf